CLINICAL TRIAL: NCT05445843
Title: KontRASt-06: An Open-label Phase II Trial Evaluating the Activity and Safety of JDQ443 Single-agent as First-line Treatment for Patients With Locally Advanced or Metastatic KRAS G12C-mutated Non-small Cell Lung Cancer With a PD-L1 Expression < 1% or a PD-L1 Expression ≥ 1% and an STK11 Co-mutation.
Brief Title: Study of Efficacy and Safety of JDQ443 Single-agent as First-line Treatment for Patients With Locally Advanced or Metastatic KRAS G12C- Mutated Non-small Cell Lung Cancer With a PD-L1 Expression < 1% or a PD-L1 Expression ≥ 1% and an STK11 Co-mutation.
Acronym: KontRASt-06
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJDQ443B12201; 2024-511708-18-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced or Metastatic KRAS G12C-mutated NSCLC With a PD-L1 Expression <1% or a PD-L1 Expression ≥ 1% and an STK11 Co-mutation
Keywords: Lung cancer; NSCLC; KRAS G12C; STK11; PD-L1; JDQ443
MeSH Terms: conditions — Lung Neoplasms | interventions — JDQ443

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A- PD-L1<1% (Experimental): Participants whose tumors harbor a KRAS G12C mutation and a PD-L1 expression < 1%, regardless of STK11 mutation status.
  Interventions: Drug: JDQ443
- Cohort B- PD-L1≥ 1% and STK11 mutation (Experimental): Participants whose tumors harbor a KRAS G12C mutation, a PD-L1 expression ≥ 1% and an STK11 co-mutation.
  Interventions: Drug: JDQ443

INTERVENTIONS:
Drug: JDQ443 — JDQ443 per os (PO) 200 mg twice a day continuously

SUMMARY:
This study aims to evaluate the antitumor activity and safety of JDQ443 single-agent as first-line treatment for participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) whose tumors harbor a KRAS G12C mutation and have a PD-L1 expression < 1% (cohort A) or a PD-L1 expression ≥ 1% and an STK11 co-mutation (cohort B).

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single-arm, multicenter, phase II study evaluating the antitumor activity and safety of JDQ443 single-agent as first-line treatment for participants with locally advanced or metastatic KRAS G12C-mutated NSCLC.

The study will have 2 non-comparative cohorts that will recruit participants in parallel according to the following characteristics:

* Cohort A: participants whose tumors harbor a KRAS G12C mutation and a PD-L1 expression < 1%, regardless of STK11 mutation status.
* Cohort B: participants whose tumors harbor a KRAS G12C mutation, a PD-L1 expression ≥ 1% and an STK11 co-mutation.

The study treatment begins on Cycle 1 Day 1 (C1D1) with the first administration of JDQ443. One treatment cycle consists of 21 (±3) days.

Study completion is defined as the earliest occurrence of one of the following:

* The last participant completes last study visit (and the assessments associated with this visit have been documented and followed-up appropriately by the Investigator), dies, withdraws consent, or is lost to follow-up, whichever comes first.]
* In the event of an early study termination decision, the date of that decision.
* Another clinical study becomes available that can continue to provide JDQ443 to study participants and all participants with ongoing treatment are transferred to that clinical study.

ELIGIBILITY:
Key Inclusion criteria

* Histologically confirmed locally advanced (stage IIIb/IIIc not eligible for definitive chemoradiation or surgical resection with curative intent) or metastatic (stage IV) NSCLC without previous systemic treatment for metastatic disease. Prior (neo)adjuvant treatment with chemotherapy and/or immunotherapy, or prior radiotherapy administered sequentially or concomitantly with chemotherapy and/or immunotherapy for localized or locally advanced disease are accepted if the time between therapy completion and enrollment is > 12 months.
* Presence of a KRAS G12C mutation (all participants) and:

  * Cohort A: PD-L1 expression < 1%, regardless of STK11 mutation status
  * Cohort B: PD-L1 expression ≥ 1% and an STK11 co-mutation
* At least one measurable lesion per RECIST 1.1.
* ECOG performance status ≤ 1.
* Participants capable of swallowing study medication.

Key Exclusion criteria

* Participants whose tumors harbor an EGFR-sensitizing mutation and/or ALK rearrangement by local laboratory testing. Participants with other known druggable alterations will be excluded, if required by local guidelines
* Previous use of a KRAS G12C inhibitor or previous systemic treatment for metastatic NSCLC.
* A medical condition that results in increased photosensitivity (i.e., solar urticaria, lupus erythematosus, etc.).
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Participants who are taking a prohibited medication (strong CYP3A inducers) that cannot be discontinued at least seven days prior to the first dose of study treatment and for the duration of the study.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- The Brown University Oncology Group, Providence, Rhode Island, United States
- Argentina (3):
  - Novartis Investigative Site, Pilar, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Austria (2):
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Wels
- Belgium (2):
  - Novartis Investigative Site, Sint-Niklaas, Oost Vlaanderen
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte
  - Novartis Investigative Site, Rio de Janeiro
- China (3):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Beijing
- France (5):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
- Germany (5):
  - Novartis Investigative Site, Kempten (Allgäu), Bavaria
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Athens, Greece
- Novartis Investigative Site, Mátraháza, Hungary
- India (2):
  - Novartis Investigative Site, Thellakom Kottayam, Kerala
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
- Italy (4):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
- Malaysia (2):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
- Netherlands (2):
  - Novartis Investigative Site, Breda, North Brabant
  - Novartis Investigative Site, Leeuwarden, Provincie Friesland
- Novartis Investigative Site, Porto, Portugal
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, Bagcilar
  - Novartis Investigative Site, Diyarbakır, Sur
  - Novartis Investigative Site, Ankara, Yenimahalle
- Novartis Investigative Site, Torquay, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted globally across 19 countries.
Groups:
- Cohort A- PD-L1<1%: Participants whose tumors harbored a KRAS G12C mutation and a PD-L1 expression < 1%, regardless of STK11 mutation status.
- Cohort B- PD-L1≥ 1% and STK11 Mutation: Participants whose tumors harbored a KRAS G12C mutation, a PD-L1 expression ≥ 1%, and an STK11 co-mutation.
Period: Overall Study
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Started (All enrolled participants were included in the Full Analysis Set (FAS) and Safety Set (SAF)) | 72 | 23
Pharmacokinetic Analysis Set (PAS) (All participants who received at least one planned dose of study treatment and provided an evaluable pharmacokinetic concentration.) | 69 | 23
Full Pharmacokinetic Analysis Set (FPAS) (PAS participants with intensive PK collection schedule who provided an evaluable PK profile.) | 14 | 9
Treatment Ongoing (Treatment ongoing at the time of the Primary Analysis data cut-off date 04-Nov-2024) | 25 | 5
Discontinued From Treatment and Continued in the Follow-up Period | 32 | 10
Discontinued From Treatment and Did Not Enter the Follow-up Period | 15 | 8
Completed | 0 | 0
Not Completed | 72 | 23
Not completed — Treatment ongoing at the time of the data cut-off date 04NOV2024 | 25 | 5
Not completed — Progressive disease | 17 | 9
Not completed — Physician Decision | 16 | 4
Not completed — Death | 6 | 3
Not completed — Subject decision | 6 | 2
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation | Total
Number analyzed (Participants) | 72 | 23 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (7.68) | 63.7 (10.29) | 66.7 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 5 | 30
  Male | 47 | 18 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 13 | 70
  Asian | 11 | 7 | 18
  Unknown | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Determined by the Investigator in Cohort A
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as best overall response (BOR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by the Investigator in Cohort A.
Time Frame: Up to approximately 22 months
Population: Full Analysis Set (FAS) comprised all participants to whom study treatment had been assigned and who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage (%) of participants
Arm/Group | Cohort A- PD-L1<1%
Number analyzed (Participants) | 72
Percentage (%) of participants | 29.2 [19.0 to 41.1]

2. Secondary Outcome: Key Secondary Outcome Measure: Overall Response Rate (ORR) as Determined by the Investigator in Cohort B
Description: Overall Response Rate (ORR) was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as best overall response (BOR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by the Investigator in Cohort B.
Time Frame: Up to approximately 22 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage (%) of participants
Arm/Group | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 23
Percentage (%) of participants | 21.7 [7.5 to 43.7]

3. Secondary Outcome: Number of Adverse Events and Serious Adverse Events as Assessed by CTCAE Criteria
Description: The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs), through the monitoring of relevant clinical and laboratory safety parameters.
  Treatment-emergent Adverse Events (TEAEs) in this study are defined as events that begin after the first dose of study treatment and continue until 30 days after the last dose of study treatment, or events that are present prior to the first dose of treatment and increase in severity based on preferred term within 30 days after the last study treatment.
Time Frame: Up to approximately 59 months
Reporting Status: Not Posted, anticipated posting 2028-11

4. Secondary Outcome: Plasma JDQ443 Concentration in All Participants
Description: JDQ443 concentration data of all participants were reported separately for each of the two cohorts and summarized using descriptive statistics.
Time Frame: Cycle 1 Day 1 (predose/0hour, 4 hours and 6 hours), Cycle 1 Day 15 (predose/0hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours and 12 hours). Cycles 3, 5 and 7 Day 1 (predose/0hour). 1 cycle = 21 days.
Population: Pharmacokinetic Analysis Set (PAS) - Participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 65 | 22
ng/mL
  Cycle 1 Day 1 (predose/0hour) | 0 (0) | 0 (0)
  Cycle 1 Day 1 (4 hours): number analyzed (Participants) | 62 | 19
  Cycle 1 Day 1 (4 hours) | 3170 (80.8) | 4980 (59.8)
  Cycle 1 Day 1 (6 hours): number analyzed (Participants) | 61 | 20
  Cycle 1 Day 1 (6 hours) | 2970 (65.6) | 4190 (65.7)
  Cycle 1 Day 15 (predose/0hour): number analyzed (Participants) | 64 | 21
  Cycle 1 Day 15 (predose/0hour) | 1580 (96.8) | 1490 (97.5)
  Cycle 1 Day 15 (1 hour): number analyzed (Participants) | 13 | 8
  Cycle 1 Day 15 (1 hour) | 2440 (102.0) | 3390 (89.3)
  Cycle 1 Day 15 (2 hours): number analyzed (Participants) | 12 | 8
  Cycle 1 Day 15 (2 hours) | 3290 (82.7) | 4700 (81.8)
  Cycle 1 Day 15 (3 hours): number analyzed (Participants) | 12 | 8
  Cycle 1 Day 15 (3 hours) | 3770 (70.4) | 5540 (41.7)
  Cycle 1 Day 15 (4 hours): number analyzed (Participants) | 60 | 18
  Cycle 1 Day 15 (4 hours) | 3290 (61.0) | 4330 (54.5)
  Cycle 1 Day 15 (6 hours): number analyzed (Participants) | 60 | 19
  Cycle 1 Day 15 (6 hours) | 2810 (69.7) | 3600 (59.9)
  Cycle 1 Day 15 (8 hours): number analyzed (Participants) | 11 | 8
  Cycle 1 Day 15 (8 hours) | 2260 (92.9) | 3120 (55.4)
  Cycle 1 Day 15 (12 hours): number analyzed (Participants) | 11 | 8
  Cycle 1 Day 15 (12 hours) | 1780 (120.5) | 2380 (72.7)
  Cycle 3 Day 1 (predose/0hour): number analyzed (Participants) | 40 | 15
  Cycle 3 Day 1 (predose/0hour) | 1060 (160.9) | 1090 (178.0)
  Cycle 5 Day 1 (predose/0hour): number analyzed (Participants) | 32 | 14
  Cycle 5 Day 1 (predose/0hour) | 1000 (73.6) | 1320 (118.4)
  Cycle 7 Day 1 (predose/0hour): number analyzed (Participants) | 33 | 12
  Cycle 7 Day 1 (predose/0hour) | 948 (74.2) | 1400 (99.4)

5. Secondary Outcome: Plasma JDQ443 Concentration in Chinese Participants
Description: JDQ443 concentration data of Chinese participants were reported separately for each of the two cohorts and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Pharmacokinetic Analysis Set (PAS) - Chinese participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 7 | 5
ng/mL
  Cycle 1 Day 1 (predose/0hour) | 0 (0) | 0 (0)
  Cycle 1 Day 1 (4 hours): number analyzed (Participants) | 7 | 4
  Cycle 1 Day 1 (4 hours) | 3480 (41.1) | 2890 (110.9)
  Cycle 1 Day 1 (6 hours) | 3220 (26.7) | 2730 (92.7)
  Cycle 1 Day 15 (predose/0hour): number analyzed (Participants) | 6 | 5
  Cycle 1 Day 15 (predose/0hour) | 1670 (95.7) | 1410 (113.8)
  Cycle 1 Day 15 (1 hour): number analyzed (Participants) | 2 | 2
  Cycle 1 Day 15 (1 hour) | 2650 (164.1) | 1470 (249.7)
  Cycle 1 Day 15 (2 hours): number analyzed (Participants) | 2 | 2
  Cycle 1 Day 15 (2 hours) | 3400 (92.3) | 2330 (252.3)
  Cycle 1 Day 15 (3 hours): number analyzed (Participants) | 2 | 2
  Cycle 1 Day 15 (3 hours) | 5390 (106.9) | 4120 (92.0)
  Cycle 1 Day 15 (4 hours): number analyzed (Participants) | 6 | 5
  Cycle 1 Day 15 (4 hours) | 3130 (114.6) | 3130 (95.2)
  Cycle 1 Day 15 (6 hours): number analyzed (Participants) | 6 | 5
  Cycle 1 Day 15 (6 hours) | 2830 (112.6) | 2670 (97.3)
  Cycle 1 Day 15 (8 hours): number analyzed (Participants) | 2 | 2
  Cycle 1 Day 15 (8 hours) | 4410 (74.8) | 2630 (133.1)
  Cycle 1 Day 15 (12 hours): number analyzed (Participants) | 2 | 2
  Cycle 1 Day 15 (12 hours) | 4290 (53.4) | 2600 (164.4)
  Cycle 3 Day 1 (predose/0hour): number analyzed (Participants) | 4 | 5
  Cycle 3 Day 1 (predose/0hour) | 1110 (42.4) | 949 (142.6)
  Cycle 5 Day 1 (predose/0hour): number analyzed (Participants) | 2 | 5
  Cycle 5 Day 1 (predose/0hour) | 650 (42.9) | 1050 (174.6)
  Cycle 7 Day 1 (predose/0hour): number analyzed (Participants) | 2 | 4
  Cycle 7 Day 1 (predose/0hour) | 1530 (60.9) | 1150 (181.6)

6. Secondary Outcome: Plasma JDQ443 Concentration in Non-Chinese Participants
Description: JDQ443 concentration data of non-Chinese participants were reported separately for each of the two cohorts and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Pharmacokinetic Analysis Set (PAS) - Non-Chinese participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 58 | 17
ng/mL
  Cycle 1 Day 1 (predose/0hour) | 0 (0) | 0 (0)
  Cycle 1 Day 1 (4 hours): number analyzed (Participants) | 55 | 15
  Cycle 1 Day 1 (4 hours) | 3140 (85.5) | 5760 (34.9)
  Cycle 1 Day 1 (6 hours): number analyzed (Participants) | 54 | 15
  Cycle 1 Day 1 (6 hours) | 2940 (69.8) | 4840 (49.9)
  Cycle 1 Day 15 (predose/0hour): number analyzed (Participants) | 58 | 16
  Cycle 1 Day 15 (predose/0hour) | 1570 (98.1) | 1510 (97.5)
  Cycle 1 Day 15 (1 hour): number analyzed (Participants) | 11 | 6
  Cycle 1 Day 15 (1 hour) | 2400 (103.1) | 4480 (23.1)
  Cycle 1 Day 15 (2 hours): number analyzed (Participants) | 10 | 6
  Cycle 1 Day 15 (2 hours) | 3270 (87.4) | 5930 (23.8)
  Cycle 1 Day 15 (3 hours): number analyzed (Participants) | 10 | 6
  Cycle 1 Day 15 (3 hours) | 3500 (67.2) | 6120 (23.9)
  Cycle 1 Day 15 (4 hours): number analyzed (Participants) | 54 | 13
  Cycle 1 Day 15 (4 hours) | 3300 (55.9) | 4910 (31.2)
  Cycle 1 Day 15 (6 hours): number analyzed (Participants) | 54 | 14
  Cycle 1 Day 15 (6 hours) | 2810 (66.2) | 4010 (43.4)
  Cycle 1 Day 15 (8 hours): number analyzed (Participants) | 9 | 6
  Cycle 1 Day 15 (8 hours) | 1950 (89.4) | 3300 (41.00)
  Cycle 1 Day 15 (12 hours): number analyzed (Participants) | 9 | 6
  Cycle 1 Day 15 (12 hours) | 1460 (116.0) | 2320 (62.3)
  Cycle 3 Day 1 (predose/0hour): number analyzed (Participants) | 36 | 10
  Cycle 3 Day 1 (predose/0hour) | 1050 (175.9) | 1180 (217.6)
  Cycle 5 Day 1 (predose/0hour): number analyzed (Participants) | 30 | 9
  Cycle 5 Day 1 (predose/0hour) | 1030 (74.7) | 1550 (90.5)
  Cycle 7 Day 1 (predose/0hour): number analyzed (Participants) | 31 | 8
  Cycle 7 Day 1 (predose/0hour) | 917 (74.4) | 1500 (85.1)

7. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) of JDQ443
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. Cmax was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 14 | 9
ng/mL
  All participants | 4170 (59.8) | 5160 (52.4)
  Chinese participants: number analyzed (Participants) | 2 | 2
  Chinese participants | 6010 (82.5) | 4320 (103.0)
  non-Chinese participants: number analyzed (Participants) | 12 | 7
  non-Chinese participants | 3920 (57.5) | 5430 (45.7)

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of JDQ443
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. Tmax was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 14 | 9
Hours
  All participants | 2.96 [0.967 to 9.50] | 3.00 [1.00 to 10.8]
  Chinese participants: number analyzed (Participants) | 2 | 2
  Chinese participants | 3.58 [3.05 to 4.10] | 3.61 [3.13 to 4.08]
  non-Chinese participants: number analyzed (Participants) | 12 | 7
  non-Chinese participants | 2.61 [0.967 to 9.50] | 2.98 [1.00 to 10.8]

9. Secondary Outcome: Time to Last Nonzero Plasma Concentration (Tlast) of JDQ443
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. Tlast was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 14 | 9
Hours
  All participants | 10.1 [6.00 to 16.9] | 11.1 [10.0 to 21.0]
  Chinese participants: number analyzed (Participants) | 2 | 2
  Chinese participants | 11.9 [11.6 to 12.2] | 11.2 [11.1 to 11.4]
  non-Chinese participants: number analyzed (Participants) | 12 | 7
  non-Chinese participants | 10.1 [6.00 to 16.9] | 11.0 [10.0 to 21.0]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞) of JDQ443
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. AUC∞ was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 3 | 2
hr*ng/mL
  All participants | 33400 (69.0) | 41800 (21.7)
  Chinese participants: number analyzed (Participants) | 0 | 0
  non-Chinese participants | 33400 (69.0) | 41800 (21.7)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Measurable Concentration (AUClast) of JDQ443
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. AUClast was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 14 | 9
hr*ng/mL
  All participants | 29100 (79.3) | 44200 (47.6)
  Chinese participants: number analyzed (Participants) | 2 | 2
  Chinese participants | 52700 (84.7) | 33500 (137.2)
  non-Chinese participants: number analyzed (Participants) | 12 | 7
  non-Chinese participants | 26400 (75.7) | 47900 (25.5)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve During a Dosage Interval (AUCτ) of JDQ443
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. AUCτ was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 12 | 9
hr*ng/mL
  All participants | 34500 (69.4) | 42700 (50.6)
  Chinese participants: number analyzed (Participants) | 2 | 2
  Chinese participants | 53500 (79.2) | 35400 (135.1)
  non-Chinese participants: number analyzed (Participants) | 10 | 7
  non-Chinese participants | 31600 (67.4) | 45100 (35.0)

13. Secondary Outcome: Total Body Clearance (CL/F) of JDQ443 in Plasma
Description: Pharmacokinetic (PK) parameters were calculated based on JDQ443 plasma concentrations and actual sampling time points. PK parameters were reported separately for all participants, non-Chinese participants, and Chinese participants in each of the two cohorts. CL/F was listed and summarized using descriptive statistics.
Time Frame: as for outcome 4
Population: Full Pharmacokinetic Analysis Set (FPAS) - Participants with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
Number analyzed (Participants) | 12 | 9
mL/hr
  All participants | 5800 (69.4) | 4680 (50.6)
  Chinese participants: number analyzed (Participants) | 2 | 2
  Chinese participants | 3730 (79.2) | 5650 (135.1)
  non-Chinese participants: number analyzed (Participants) | 10 | 7
  non-Chinese participants | 6340 (67.4) | 4440 (35.0)

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to the cut-off date for the primary analysis (04-Nov-2024), approximately 22 months.
Arm/Group | Cohort A- PD-L1<1% | Cohort B- PD-L1≥ 1% and STK11 Mutation
All-Cause Mortality (participants affected / at risk) | 15/72 | 4/23
Serious Adverse Events (participants affected / at risk) | 29/72 | 10/23
Other Adverse Events (participants affected / at risk) | 60/72 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A- PD-L1<1% (N=72) | Cohort B- PD-L1≥ 1% and STK11 Mutation (N=23)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Intracranial tumour haemorrhage (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A- PD-L1<1% (N=72) | Cohort B- PD-L1≥ 1% and STK11 Mutation (N=23)
Anaemia (Blood and lymphatic system disorders) | 21 | 4
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 12 | 6
Diarrhoea (Gastrointestinal disorders) | 19 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 18 | 5
Vomiting (Gastrointestinal disorders) | 8 | 2
Asthenia (General disorders) | 14 | 3
Fatigue (General disorders) | 13 | 4
General physical health deterioration (General disorders) | 0 | 3
Oedema (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 13 | 5
Pyrexia (General disorders) | 8 | 3
Pneumonia (Infections and infestations) | 4 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Alanine aminotransferase increased (Investigations) | 5 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 4
Blood creatinine increased (Investigations) | 6 | 1
Blood magnesium decreased (Investigations) | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 2
Weight decreased (Investigations) | 8 | 5
White blood cell count decreased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 5 | 3
Insomnia (Psychiatric disorders) | 5 | 0
Haematuria (Renal and urinary disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 4
Hypotension (Vascular disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT05445843/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT05445843/SAP_001.pdf